CLINICAL TRIAL: NCT07310680
Title: Impact of mHealth Education on Hemoglobin Level Among Pregnant Women With Anemia in Rural Bangladesh.
Acronym: Mobile Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: North South University, Bangladesh (Unknown)
Responsible Party: Principal Investigator, Ananta Taiyaba Tabassum, Doctoral Student (PhD), Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: #2025/OR-NSU/IRB/0917
Record Dates: First submitted 2025-11-24; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Anemia; Pregnant Women
Keywords: Anemia; Pregnant women; mHealth; Bangladesh
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile health education intervention (Experimental): mHealth education intervention to increase hemoglobin level in pregnancy
  Interventions: Other: mHealth education
- Usual care: Control group (No Intervention): No mHealth education: Usual care

INTERVENTIONS:
Other: mHealth education — Mobile health education to increase hemoglobin level among pregnant women
  Arms: Mobile health education intervention

SUMMARY:
Anemia in pregnancy can result in negative pregnancy outcomes, which are higher among pregnant women of rural Bangladesh. A cost-effective health education program is urgently needed to introduce, which will help to improve their hemoglobin level by changing their lifestyle. In many rural settings, mobile-based health (mHealth) education programs have been shown to improve hemoglobin levels effectively during the antenatal period. So, we aim to assess the impact of a mHealth education program on improving hemoglobin levels among anemic pregnant women of rural Bangladesh.

The study will be carried out in the rural settings of a district of Bangladesh named Chandpur. This study timeline is from December 2025 to May 2026.

After this survey, a randomized controlled trial study will be conducted where 160 pregnant women who are diagnosed with mild and moderate anemia will be offered to participate. Pregnant women who will give informed consent will be randomly assigned to two arms: intervention and control. Every arm will have an equal number of anemic pregnant women. Pregnant women in the intervention arm will receive anemia management-related health education through mobile messages and calls. This intervention program will educate pregnant women about the causes, risks, and symptoms of anemia, with the prevention strategies like dietary improvement, supplementation, parasitic disease control, safe motherhood, family planning, and iron-rich food production. Additionally, they will get regular care, a booklet and reminders of ANC visits during the study period. In contrast, the pregnant women of the control arm will receive regular care during this period, but after the end-line assessment, they will also get the booklet. After 4 months of the intervention program, the end-line assessment will be done, where the hemoglobin, nutritional status, and literacy about anemia will be assessed. Multiple comparisons will be performed by two-way analysis of variance tests for the evaluation of the outcome variables. Additionally, a Generalized Estimating Equations (GEE) model will be used to analyze the effect of the mHealth education program on related factors. A p-value less than 0.5 will be considered significant in this study.

If this mHealth-based education program shows improvement in hemoglobin level, this can be utilized in low-resource settings widely to ensure safe pregnancy outcomes in the future.

DETAILED DESCRIPTION:
Anemia is a public health problem in which the hemoglobin level becomes lower than the recommended value of 11.0 grams per deciliter (gm/dl) in blood. Generally, pregnant women are more vulnerable to developing anemia due to increased physiological demand for their growing fetus. In pregnancy, a low iron store is the most common cause of low hemoglobin levels, and therefore, 27 milligrams (mg) of oral iron needs to be taken daily during this period. A pregnant woman with anemia can experience fatigue, cold, shortness of breath, dizziness, headache, a fast heartbeat, restless leg syndrome, and so on. If this condition is untreated, adverse events can occur, such as preeclampsia, fatigue, hypertensive disorders, intrauterine growth restriction, placental abnormalities, threatened abortion, emotional disturbances, increased susceptibility to infections, poor weight gain, and preterm labor, which usually later lead to maternal or neonatal death.

Anemia during pregnancy is responsible for about 20% of maternal deaths per year, and globally its prevalence is 40.05%, including 42.7% in low- and middle-income countries (LMICs). The prevalence of anemia in South Asian countries is also alarming, and the rate of decline has been notably slow. Since the majority of the population in this region resides in rural areas, low literacy levels and poor financial conditions have led to limited access to proper healthcare. The long-term effect of gestational anemia is a loss of human productivity, which is one actual reason for the slow economic development in these regions. Like Nepal (43.1%), Pakistan (57.7%), and India (52.2%), Bangladesh is also noted to have a high prevalence (50%) of anemia among rural pregnant women. Unawareness about anemia, poverty, inadequate nutrition, early marriage, improper dietary practice, low educational qualification, women's unemployment, women's inequality, low access to health care facilities, low supplement compliance, and not visiting antenatal care (ANC) are the underlying factors of anemia among Bangladeshi pregnant women.

To control this issue, an effective intervention program is urgently needed to be implemented in this region. There are numerous programs available; however, educational intervention programs have been proven effective in these types of rural and low-resource settings. Usually, in these educational intervention programs, rural pregnant women are introduced to anemia, its symptoms, cause, consequences, when to see a doctor, how to manage this, effective preventive measures including Iron and Folic Acid (IFA) supplements, proper hygiene, dietary knowledge, and other things related to anemia reduction. By improving their lifestyle and awareness of anemia, this information ultimately helps them raise their hemoglobin level during pregnancy.

In Bangladesh, several educational intervention programs have been implemented previously; however, the national prevalence rate remains higher, with a target of being controlled under 25% by 2025. Until now, education programs in Bangladesh have been carried out at the community level or through a handbook. However, in these programs, factors such as forgetfulness, transportation issues, feeling weak, bad weather, inability to read, and being preoccupied with family are reported as causes of participant loss and program failure. Furthermore, the majority of them seek to reduce maternal risks among pregnant women by providing general maternal-related health information, but an educational intervention study solely focused on anemia in pregnancy has not been identified in Bangladesh.

In this digital technology era, using the telecommunication method to provide education-based intervention programs is expected to improve not only the accessibility of proper information on anemia management at the individual level but also affordability for the participants. Mobile-based Health (mHealth) education programs on anemia in pregnancy have been introduced in many other countries like Malaysia, Saudi Arabia, Ethiopia, and Nepal as an intervention. In these programs, voice calls, text, and/or audio messages through personal mobile phones have been used to deliver educational information to pregnant women. Moreover, in those studies, mHealth has given better results in increasing hemoglobin levels in pregnant women than many other conventional treatments. According to the Bangladesh Demographic Health Survey (BDHS) 2022 report, approximately 98% of the total population and 68% of rural married women aged between 15-49 years own at least one mobile phone in Bangladesh. In addition, a previous study confirmed that using a mobile phone for pregnancy-related purposes has a positive relation with mothers' receipt of antenatal care in Bangladesh. Therefore, we should seize this opportunity to strengthen maternal healthcare and evaluate mHealth-based education for improving hemoglobin levels in anemic pregnant women, an area yet to be studied. Due to this existing gap and need, this study aims to evaluate the impact of mHealth education on anemia, specifically focusing on its effectiveness in increasing hemoglobin levels among anemic pregnant women in rural areas of Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

- 1. Pregnant women who will be diagnosed with mild and moderate anemia (Blood hemoglobin levels are between 7g/dL and 10.9 g/dL).

2. Have at least one active mobile phone in the family. 3. Those who will give written informed consent to participate in the intervention study at the time of enrollment

Exclusion Criteria:

- 1. Hospitalized at the time of the study period. 2. Women with any known or suspected chronic or congenital disease, such as blood inflammation, diabetic mellitus, thalassemia, hypertension, and psychiatric illness.

3. Those who have severe anemia. 4. Having the possibility of leaving the study area during this study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 132 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of mHealth education intervention with changes in blood hemoglobin level | 4 months
  Individual pregnant women will have their anemia status assessed (non-anemic, mild, moderate, and severe anemia) based on blood hemoglobin measurement using an automated hematology analyzer. According to the World Health Organization (WHO), hemoglobin levels <11.0 g/dL will be considered indicative of anemia among pregnant women. Hemoglobin concentrations of 10.0-10.9 g/dL, 7.0-9.9 g/dL, and <7.0 g/dL will be classified as mild, moderate, and severe anemia, respectively, while hemoglobin levels ≥11.0 g/dL will be considered non-anemic.
  Following the mHealth education intervention, changes in anemia status will be assessed from baseline to endline among pregnant women, including transitions from anemic to non-anemic, severe to moderate/mild/non-anemic, moderate to mild/non-anemic, and mild to non-anemic, in both the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yoko Shimpuku, RN PhD, Study Director — Graduate School of Biomedical and Health Sciences, Hiroshima university
Locations (1):
- Upazilla Health Complex and Community Clinic, Chāndpur, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Due to ethical constraints, the IPD will be securely stored and will not be shared with researchers outside the primary research team.